CLINICAL TRIAL: NCT01768559
Title: A Randomized, Open-label, Active-controlled, 3-arm Parallel-group, 26-week Study Comparing the Efficacy and Safety of Lixisenatide to That of Insulin Glulisine Once Daily and Insulin Glulisine Three Times Daily in Patients With Type 2 Diabetes Insufficiently Controlled With Insulin Glargine With or Without Metformin
Brief Title: Efficacy and Safety of Lixisenatide Versus Insulin Glulisine on Top of Insulin Glargine With or Without Metformin in Type 2 Diabetic Patients
Acronym: GetGoal-Duo-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC12626; 2012-004096-38 (EudraCT Number); U1111-1131-4936 (Other: UTN)
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Insulin Glargine; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lixisenatide (Experimental): Lixisenatide 10 mcg once daily (QD) for 2 weeks post-randomization, then at a maintenance dose of 20 mcg QD up to Week 26 on top of insulin glargine with or without metformin.
  Interventions: Drug: Lixisenatide (AVE0010); Drug: Insulin Glargine (Mandatory background drug); Drug: Metformin (Background drug)
- Insulin Glulisine QD (Active Comparator): Insulin glulisine QD from randomization up to Week 26 on top of Insulin glargine with or without metformin.
  Interventions: Drug: Insulin glulisine QD; Drug: Insulin Glargine (Mandatory background drug); Drug: Metformin (Background drug)
- Insulin Glulisine TID (Active Comparator): Insulin glulisine thrice daily (TID) from randomization up to Week 26 on top of Insulin glargine with or without metformin.
  Interventions: Drug: Insulin glulisine TID; Drug: Insulin Glargine (Mandatory background drug); Drug: Metformin (Background drug)

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Pharmaceutical form: Solution for injection; Route of administration: Self-administered by subcutaneous injection 30 to 60 minutes before breakfast or dinner.
  Other Names: Lyxumia®; Device: Disposable self-injector prefilled pen (Delta 14®)
  Arms: Lixisenatide
Drug: Insulin glulisine QD — Pharmaceutical form: Solution for injection; Route of administration: Self-administered by subcutaneous injection within 15 minutes before breakfast or dinner. The initial dose was 3-5 units and then individually titrated to obtain the SMPG value >5.6 mmol/L (100 mg/dL) and ≤7.8 mmol/L (140 mg/dL) before lunch (if administered at breakfast) or at bedtime (if administered at dinner).
  Other Names: HMR1964; Device: Disposable self-injector prefilled pen (Apidra® Solostar®)
  Arms: Insulin Glulisine QD
Drug: Insulin glulisine TID — Pharmaceutical form: Solution for injection; Route of administration: Self-administered by subcutaneous injection within 15 minutes before each meal. The initial dose was 3-5 units for each meal and then individually titrated to obtain the SMPG value >5.6 mmol/L (100 mg/dL) and ≤7.8 mmol/L (140 mg/dL) before the next meal or at bedtime (for injection at dinner).
  Other Names: HMR1964; Device: Disposable self-injector prefilled pen (Apidra® Solostar®)
  Arms: Insulin Glulisine TID
Drug: Insulin Glargine (Mandatory background drug) — Pharmaceutical form: Solution for injection; Route of administration: Self-administered by subcutaneous injection at breakfast or dinner. Doses were adjusted to maintain a fasting self-monitored plasma glucose (SMPG) between 4.4 to 5.6 mmol/L (80 to 100 mg/dL).
  Other Names: Device: Disposable self-injector prefilled pen (Lantus® Solostar®)
Drug: Metformin (Background drug) — Pharmaceutical form: Tablet; Route of administration: Oral administration. If previously taken, Metformin to be continued at stable dose (≥1.5 g/day) throughout the study.

SUMMARY:
Primary Objective:

- To compare lixisenatide versus insulin glulisine in terms of glycosylated hemoglobin (HbA1c) reduction and body weight change at Week 26 in type 2 diabetic participants not adequately controlled on insulin glargine ± metformin.

Secondary Objectives:

- To compare the treatments/regimens on:

* The percentage of participants reaching the target of HbA1c <7% or ≤6.5%,
* Body weight,
* Self-Monitored Glucose profiles,
* Fasting Plasma Glucose (FPG),
* Post-prandial plasma glucose (PPG) /glucose excursions during a standardized meal test (subset of participants),
* Daily doses of insulins,
* Safety and tolerability.

DETAILED DESCRIPTION:
Approximately 41 weeks including a 26 week treatment period.

ELIGIBILITY:
Inclusion criteria :

* Participants with type 2 diabetes mellitus diagnosed at least 1 year before screening visit (V1).
* Participants treated with basal insulin for at least 6 months.
* Participants treated for at least 3 months prior to visit 1 with a stable basal insulin regimen (i.e. type of insulin and time/frequency of the injection). The insulin dose should be stable (± 20%) and ≥20 U/day for at least 2 months prior to visit 1.
* Participants treated with basal insulin alone or in combination with 1 to 3 oral anti-diabetic drugs (OADs) that could be: metformin (≥1.5 g/day or maximal tolerated dose), a sulfonylurea (SU), a dipeptidyl-peptidase-4 (DPP-4) inhibitor, a glinide. The dose of OADs should be stable for at least 3 months prior to visit 1.

Exclusion criteria:

* At screening: age < legal age of majority.
* At screening, HbA1c: <7.5% and >10.0% for participants treated with basal insulin alone or in combination with metformin only; < 7.0% and > 10.0% for participants treated with basal insulin and a combination of oral anti-diabetic drugs which included a SU and/or a DPP-4 inhibitor and/or a glinide.
* Women of childbearing potential with no effective contraceptive method, pregnancy or lactation.
* Type 1 diabetes mellitus.
* Treatment with glucose-lowering agent(s) other than stated in the inclusion criteria within 3 months prior to screening.
* Previous treatment with short or rapid acting insulin other than in relation to hospitalization or an acute illness.
* Any previous treatment with lixisenatide, or any discontinuation from another glucagon-like peptide 1 (GLP-1) receptor agonist due to safety/tolerability issue or lack of efficacy.
* At screening, Body Mass Index (BMI) ≤20 or >40 kg/m^2.
* Weight change of more than 5 kg during the 3 months prior to the screening visit; use of weight loss drugs within 3 months prior to screening.
* Within the last 6 months prior to screening: history of myocardial infarction, stroke, or heart failure requiring hospitalization. Planned coronary, carotid or peripheral artery revascularisation procedures.
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery.
* At screening resting systolic blood pressure >180 mmHg or diastolic blood pressure >95 mmHg.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic condition that predisposed to MTC (e.g. multiple endocrine neoplasia syndromes).
* Contraindication related to metformin (for participant receiving this treatment), insulin glargine, insulin glulisine or lixisenatide.
* Participants with severe renal impairment (creatinine clearance less than 30 ml/min) or end-stage renal disease.
* At screening, amylase and/or lipase >3 times the upper limit of the normal laboratory range (ULN).
* At screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 ULN.
* At screening calcitonin ≥20 pg/ml (5.9 pmol/L).

Exclusion Criteria for randomization at the end of the screening period before randomization:

* HbA1c <7.0% or >9.0%.
* 7-day mean fasting SMPG >140 mg/dl (7.8 mmol/L).
* Amylase and/or lipase >3 times ULN.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 894 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (199):
- United States (46):
  - Investigational Site Number 840043, Sun City, Arizona
  - Investigational Site Number 840042, Tempe, Arizona
  - Investigational Site Number 840003, Little Rock, Arkansas
  - Investigational Site Number 840031, La Mesa, California
  - Investigational Site Number 840005, Mission Viejo, California
  - Investigational Site Number 840057, Northridge, California
  - Investigational Site Number 840035, Santa Ana, California
  - Investigational Site Number 840002, Temecula, California
  - Investigational Site Number 840037, Walnut Creek, California
  - Investigational Site Number 840023, West Hills, California
  - Investigational Site Number 840041, Denver, Colorado
  - Investigational Site Number 840012, Miami, Florida
  - Investigational Site Number 840061, Miami, Florida
  - Investigational Site Number 840045, Lawrenceville, Georgia
  - Investigational Site Number 840036, Nampa, Idaho
  - Investigational Site Number 840024, Chicago, Illinois
  - Investigational Site Number 840009, Evanston, Illinois
  - Investigational Site Number 840004, Avon, Indiana
  - Investigational Site Number 840055, Avon, Indiana
  - Investigational Site Number 840027, Des Moines, Iowa
  - Investigational Site Number 840006, Wichita, Kansas
  - Investigational Site Number 840047, Lexington, Kentucky
  - Investigational Site Number 840056, Paducah, Kentucky
  - Investigational Site Number 840022, Marrero, Louisiana
  - Investigational Site Number 840016, Baltimore, Maryland
  - Investigational Site Number 840017, Rockville, Maryland
  - Investigational Site Number 840025, Buckley, Michigan
  - Investigational Site Number 840048, Dearborn, Michigan
  - Investigational Site Number 840026, Kalamazoo, Michigan
  - Investigational Site Number 840049, Las Vegas, Nevada
  - Investigational Site Number 840029, New Hyde Park, New York
  - Investigational Site Number 840060, Smithtown, New York
  - Investigational Site Number 840030, Staten Island, New York
  - Investigational Site Number 840011, Salisbury, North Carolina
  - Investigational Site Number 840028, Fargo, North Dakota
  - Investigational Site Number 840007, Oklahoma City, Oklahoma
  - Investigational Site Number 840021, Pittsburgh, Pennsylvania
  - Investigational Site Number 840052, Myrtle Beach, South Carolina
  - Investigational Site Number 840032, Chattanooga, Tennessee
  - Investigational Site Number 840033, Nashville, Tennessee
  - Investigational Site Number 840034, Corpus Christi, Texas
  - Investigational Site Number 840001, Dallas, Texas
  - Investigational Site Number 840020, Houston, Texas
  - Investigational Site Number 840018, Norfolk, Virginia
  - Investigational Site Number 840015, Salem, Virginia
  - Investigational Site Number 840010, Milwaukee, Wisconsin
- Canada (18):
  - Investigational Site Number 124008, Brampton
  - Investigational Site Number 124015, Burlington
  - Investigational Site Number 124018, Chatham
  - Investigational Site Number 124004, Coquitlam
  - Investigational Site Number 124016, Etobicoke
  - Investigational Site Number 124014, Hamilton
  - Investigational Site Number 124020, Montreal
  - Investigational Site Number 124011, Montreal
  - Investigational Site Number 124017, Newmarket
  - Investigational Site Number 124021, Québec
  - Investigational Site Number 124003, Red Deer
  - Investigational Site Number 124012, Saint Romuald
  - Investigational Site Number 124002, Sherbrooke
  - Investigational Site Number 124001, Toronto
  - Investigational Site Number 124010, Toronto
  - Investigational Site Number 124005, Vancouver
  - Investigational Site Number 124006, Victoria
  - Investigational Site Number 124007, Winnipeg
- Chile (8):
  - Investigational Site Number 152103, Santiago
  - Investigational Site Number 152107, Santiago
  - Investigational Site Number 152101, Santiago
  - Investigational Site Number 152105, Santiago
  - Investigational Site Number 152102, Santiago
  - Investigational Site Number 152106, Santiago
  - Investigational Site Number 152108, Santiago
  - Investigational Site Number 152109, Santiago
- Czechia (8):
  - Investigational Site Number 203107, Beroun
  - Investigational Site Number 203103, Jílové u Prahy
  - Investigational Site Number 203101, Ostrava
  - Investigational Site Number 203110, Police nad Metují
  - Investigational Site Number 203105, Prague
  - Investigational Site Number 203102, Prague
  - Investigational Site Number 203108, Prague
  - Investigational Site Number 203104, Trutnov
- Estonia (4):
  - Investigational Site Number 233102, Pärnu
  - Investigational Site Number 233103, Tallinn
  - Investigational Site Number 233104, Tallinn
  - Investigational Site Number 233101, Viljandimaa
- France (9):
  - Investigational Site Number 250108, Bois-Guillaume
  - Investigational Site Number 250105, Corbeil-Essonnes
  - Investigational Site Number 250104, La Rochelle
  - Investigational Site Number 250106, Lyon
  - Investigational Site Number 250107, Lyon
  - Investigational Site Number 250109, Mantes-la-Jolie
  - Investigational Site Number 250102, Paris
  - Investigational Site Number 250101, Vandœuvre-lès-Nancy
  - Investigational Site Number 250103, Vénissieux
- Germany (13):
  - Investigational Site Number 276112, Bad Mergentheim
  - Investigational Site Number 276108, Berlin
  - Investigational Site Number 276102, Dortmund
  - Investigational Site Number 276120, Dresden
  - Investigational Site Number 276106, Dresden
  - Investigational Site Number 276117, Frankfurt A.M.
  - Investigational Site Number 276116, Görlitz
  - Investigational Site Number 276113, Heidelberg
  - Investigational Site Number 276118, Leipzig
  - Investigational Site Number 276119, Magdeburg
  - Investigational Site Number 276103, Neumünster
  - Investigational Site Number 276109, Saint Ingbert-Oberwürzbach
  - Investigational Site Number 276115, Speyer
- Hungary (8):
  - Investigational Site Number 348107, Budapest
  - Investigational Site Number 348108, Budapest
  - Investigational Site Number 348102, Budapest
  - Investigational Site Number 348101, Eger
  - Investigational Site Number 348103, Pápa
  - Investigational Site Number 348106, Sátoraljaújhely
  - Investigational Site Number 348104, Szeged
  - Investigational Site Number 348105, Zalaegerszeg
- Italy (5):
  - Investigational Site Number 380103, Bologna
  - Investigational Site Number 380102, Catania
  - Investigational Site Number 380101, Milan
  - Investigational Site Number 380105, Napoli
  - Investigational Site Number 380104, Torino
- Latvia (5):
  - Investigational Site Number 428103, Jelgava
  - Investigational Site Number 428104, Ogre
  - Investigational Site Number 428102, Riga
  - Investigational Site Number 428105, Riga
  - Investigational Site Number 428101, Sigulda
- Lithuania (5):
  - Investigational Site Number 440104, Jonava
  - Investigational Site Number 440103, Kaunas
  - Investigational Site Number 440102, Kaunas
  - Investigational Site Number 440101, Kaunas
  - Investigational Site Number 440105, Klaipėda
- Mexico (11):
  - Investigational Site Number 484108, Chihuahua City
  - Investigational Site Number 484101, Cuernavaca
  - Investigational Site Number 484111, Durango
  - Investigational Site Number 484104, Guadalajara
  - Investigational Site Number 484109, Guadalajara
  - Investigational Site Number 484107, Guadalajara
  - Investigational Site Number 484105, Guadalajara
  - Investigational Site Number 484110, Guadalajara
  - Investigational Site Number 484103, Mexico City
  - Investigational Site Number 484102, México
  - Investigational Site Number 484106, Monterrey
- Poland (7):
  - Investigational Site Number 616101, Bialystok
  - Investigational Site Number 616103, Bydgoszcz
  - Investigational Site Number 616102, Bytom
  - Investigational Site Number 616106, Krakow
  - Investigational Site Number 616104, Krakow
  - Investigational Site Number 616105, Puławy
  - Investigational Site Number 616107, Warsaw
- Romania (17):
  - Investigational Site Number 642105, Bacau
  - Investigational Site Number 642108, Cluj-Napoca
  - Investigational Site Number 642106, Deva
  - Investigational Site Number 642113, Galati
  - Investigational Site Number 642107, Hunedoara
  - Investigational Site Number 642117, Iași
  - Investigational Site Number 642103, Oradea
  - Investigational Site Number 642104, Oradea
  - Investigational Site Number 642112, Piteşti
  - Investigational Site Number 642114, Ploieşti
  - Investigational Site Number 642102, Reşiţa
  - Investigational Site Number 642111, Sibiu
  - Investigational Site Number 642109, Târgu Mureş
  - Investigational Site Number 642110, Târgu Mureş
  - Investigational Site Number 642116, Timișoara
  - Investigational Site Number 642101, Timișoara
  - Investigational Site Number 642115, Timișoara
- Russia (11):
  - Investigational Site Number 643111, Moscow
  - Investigational Site Number 643107, Moscow
  - Investigational Site Number 643105, Moscow
  - Investigational Site Number 643110, Penza
  - Investigational Site Number 643101, Saint Petersburg
  - Investigational Site Number 643104, Saint Petersburg
  - Investigational Site Number 643109, Saint Petersburg
  - Investigational Site Number 643106, Saint Petersburg
  - Investigational Site Number 643108, Saint Petersburg
  - Investigational Site Number 643103, Saint Petersburg
  - Investigational Site Number 643102, Saratov
- Spain (4):
  - Investigational Site Number 724105, A Coruña
  - Investigational Site Number 724102, Ferrol
  - Investigational Site Number 724103, Málaga
  - Investigational Site Number 724104, Seville
- Ukraine (8):
  - Investigational Site Number 804104, Chernivtsi
  - Investigational Site Number 804107, Donetsk
  - Investigational Site Number 804103, Donetsk
  - Investigational Site Number 804108, Mykolaiv
  - Investigational Site Number 804110, Odesa
  - Investigational Site Number 804105, Vinnytsia
  - Investigational Site Number 804102, Vinnytsia
  - Investigational Site Number 804111, Zaporizhia
- United Kingdom (12):
  - Investigational Site Number 826006, Ashton-under-Lyne
  - Investigational Site Number 826002, Birmingham
  - Investigational Site Number 826007, Carmarthen
  - Investigational Site Number 826005, Chester
  - Investigational Site Number 826008, Coventry
  - Investigational Site Number 826009, Dundee
  - Investigational Site Number 826001, Durham
  - Investigational Site Number 826011, Haddington
  - Investigational Site Number 826012, Leicester
  - Investigational Site Number 826010, Plymouth
  - Investigational Site Number 826004, Sheffield
  - Investigational Site Number 826003, St Helens

REFERENCES:
- [Result] Rosenstock J, Guerci B, Hanefeld M, Gentile S, Aronson R, Tinahones FJ, Roy-Duval C, Souhami E, Wardecki M, Ye J, Perfetti R, Heller S; GetGoal Duo-2 Trial Investigators. Prandial Options to Advance Basal Insulin Glargine Therapy: Testing Lixisenatide Plus Basal Insulin Versus Insulin Glulisine Either as Basal-Plus or Basal-Bolus in Type 2 Diabetes: The GetGoal Duo-2 Trial. Diabetes Care. 2016 Aug;39(8):1318-28. doi: 10.2337/dc16-0014. Epub 2016 May 23. PMID 27222510
- [Derived] Tabak AG, Anderson J, Aschner P, Liu M, Saremi A, Stella P, Tinahones FJ, Wysham C, Meier JJ. Efficacy and Safety of iGlarLixi, Fixed-Ratio Combination of Insulin Glargine and Lixisenatide, Compared with Basal-Bolus Regimen in Patients with Type 2 Diabetes: Propensity Score Matched Analysis. Diabetes Ther. 2020 Jan;11(1):305-318. doi: 10.1007/s13300-019-00735-7. Epub 2019 Dec 17. PMID 31848983
- [Derived] Rosenstock J, Handelsman Y, Vidal J, Ampudia Blasco FJ, Giorgino F, Liu M, Perfetti R, Meier JJ. Propensity-score-matched comparative analyses of simultaneously administered fixed-ratio insulin glargine 100 U and lixisenatide (iGlarLixi) vs sequential administration of insulin glargine and lixisenatide in uncontrolled type 2 diabetes. Diabetes Obes Metab. 2018 Dec;20(12):2821-2829. doi: 10.1111/dom.13462. Epub 2018 Aug 13. PMID 29974618

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 199 centers in 18 countries. A total of 2159 participants were screened between January 08, 2013 and April 10, 2014.
Pre-assignment Details: Participants underwent a 12-week run-in period with switch from other basal insulins to insulin glargine. A total of 1265 participants were screen failures/run-in failures; the most frequent reason for run-in failure was that glycosylated hemoglobin (HbA1c) criteria were not met at the end of run-in phase. 894 participants were randomized.
Groups:
- Lixisenatide: Lixisenatide 10 mcg once daily (QD) subcutaneously (SC) for 2 weeks, then at a maintenance dose of 20 mcg QD up to Week 26 on top of insulin glargine with or without metformin.
- Insulin Glulisine QD: Insulin glulisine QD SC up to Week 26 on top of insulin glargine with or without metformin.
- Insulin Glulisine TID: Insulin glulisine thrice daily (TID) SC up to Week 26 on top of insulin glargine with or without metformin.
Period: Overall Study
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Started | 298 | 298 | 298
Treated | 298 | 298 (1 participant received Insulin Glulisine TID (for more than 50%)) | 297 (4 participants received Insulin Glulisine QD (for more than 50%))
Completed | 268 | 281 | 285
Not Completed | 30 | 17 | 13
Not completed — Randomized but not treated | 0 | 0 | 1
Not completed — Adverse Event | 15 | 2 | 5
Not completed — Lack of Efficacy | 6 | 4 | 0
Not completed — Poor compliance to protocol | 0 | 3 | 2
Not completed — Other than specified | 9 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Lixisenatide: Lixisenatide 10 mcg QD SC for 2 weeks, then at a maintenance dose of 20 mcg QD up to Week 26 on top of insulin glargine with or without metformin.
- Insulin Glulisine TID: Insulin glulisine TID SC up to Week 26 on top of insulin glargine with or without metformin.
- Total: Total of all reporting groups
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID | Total
Number analyzed (Participants) | 298 | 298 | 298 | 894
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (8.6) | 60.2 (8.6) | 59.4 (9.5) | 59.8 (8.9)
Gender [Count of Participants; unit: Participants]
  Female | 160 | 163 | 166 | 489
  Male | 138 | 135 | 132 | 405
Race [Number; unit: participants]
  Caucasian/White | 276 | 280 | 272 | 828
  Black | 13 | 11 | 12 | 36
  Asian/Oriental | 9 | 7 | 13 | 29
  Other | 0 | 0 | 1 | 1
Ethnicity [Number; unit: participants]
  Hispanic | 63 | 58 | 68 | 189
  Non-Hispanic | 235 | 240 | 230 | 705
Metformin Use at Screening [Number; unit: participants]
  Yes | 262 | 260 | 259 | 781
  No | 36 | 38 | 39 | 113
Number of Participants with Categorical Body Mass Index (BMI) [Number; unit: participants]
  <30 kg/m^2 | 97 | 118 | 97 | 312
  ≥30 kg/m^2 | 201 | 180 | 200 | 581
  Participants not analyzed for BMI | 0 | 0 | 1 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] — 893 participants (298 in Lixisenatide arm; 298 in Insulin glulisine QD and 297 in Insulin glulisine TID) were included for baseline BMI analysis.
  kg/m^2 | 32.27 (4.57) | 31.86 (4.39) | 32.50 (4.60) | 32.21 (4.52)
Weight [Mean (Standard Deviation); unit: kg] — 893 participants (298 in Lixisenatide arm, 298 in Insulin glulisine QD and 297 in Insulin glulisine TID) were included for baseline weight analysis.
  kg | 90.06 (17.31) | 88.45 (15.84) | 90.08 (17.18) | 89.53 (16.79)
HbA1c [Mean (Standard Deviation); unit: percentage of hemoglobin] — 893 participants (298 in Lixisenatide arm; 298 in Insulin glulisine QD and 297 in Insulin glulisine TID) were included for HbA1c analysis.
  percentage of hemoglobin | 7.77 (0.55) | 7.73 (0.59) | 7.79 (0.60) | 7.76 (0.58)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] — 893 participants (298 in Lixisenatide arm; 298 in Insulin glulisine QD and 297 in Insulin glulisine TID) were included for FPG analysis.
  mmol/L | 6.58 (1.82) | 6.84 (1.98) | 6.65 (1.89) | 6.69 (1.90)
2-Hour Postprandial Plasma Glucose (PPG) [Mean (Standard Deviation); unit: mmol/L] — 258 participants (79 in Lixisenatide arm; 77 in Insulin glulisine QD and 102 in Insulin glulisine TID) were included for PPG analysis.
  mmol/L | 14.26 (3.55) | 14.02 (3.59) | 14.25 (3.35) | 14.18 (3.47)
2-Hour Glucose Excursion [Mean (Standard Deviation); unit: mmol/L] — 243 participants (73 in Lixisenatide arm, 74 in Insulin glulisine QD and 96 in Insulin glulisine TID) were included for 2-hour glucose excursion analysis.
  mmol/L | 7.31 (3.19) | 7.31 (3.63) | 7.35 (3.34) | 7.33 (3.37)
Average 7-Point Self-monitored Plasma Glucose (SMPG) [Mean (Standard Deviation); unit: mmol/L] — 877 participants (292 in Lixisenatide arm; 291 in Insulin glulisine QD and 294 in Insulin glulisine TID) were included for average 7-point SMPG analysis.
  mmol/L | 9.02 (1.75) | 9.07 (1.74) | 8.99 (1.57) | 9.02 (1.68)
Insulin Glargine Dose [Mean (Standard Deviation); unit: Units (U)] — 893 participants (298 in Lixisenatide arm; 298 in Insulin glulisine QD and 297 in Insulin glulisine TID) were included for Insulin glargine dose analysis.
  Units (U) | 67.25 (31.95) | 64.72 (32.07) | 64.97 (26.90) | 65.65 (30.39)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 11.89 (6.43) | 12.33 (6.75) | 12.41 (6.80) | 12.21 (6.66)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: Change in HbA1C was calculated by subtracting baseline value from Week 26 value. Missing data was imputed using last on-treatment observation carried forward (LOCF). On-treatment period for this efficacy variable was defined as the time from the first dose of study drug up to 14 days after the last dose of study drug. Here, number of participants analyzed = participants with baseline and at least one post-baseline HbA1c assessment during on-treatment period.
Time Frame: Baseline, Week 26
Population: modified intent-to-treat (mITT) population: all randomized participants who received at least one dose of study drug; and had both baseline and at least one post-baseline efficacy assessment, irrespective of compliance with study protocol/procedures.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 292 | 292 | 295
percentage of hemoglobin | -0.63 (0.054) | -0.58 (0.054) | -0.84 (0.053)
Statistical Analysis 1: Comparison: Lixisenatide vs Insulin Glulisine QD; Analysis was performed using analysis of covariance (ANCOVA) model with treatment groups, strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of metformin use, and country as fixed effects and baseline HbA1c value as a covariate. The non-inferiority was assessed using upper bound of 2-sided 95% Confidence Interval (CI); Test type: Non-Inferiority or Equivalence — Pre-specified non-inferiority margin of 0.4%; ANCOVA; Least Square (LS) Mean Difference = -0.05, 95% CI 2-sided [-0.17 to 0.064], Standard Error of Mean 0.059 — Lixisenatide vs Insulin Glulisine QD
Statistical Analysis 2: Comparison: Lixisenatide vs Insulin Glulisine TID; Analysis was performed using ANCOVA model as described above. Hochberg procedure was used to control type 1 error at significance level = 0.025 (1-sided) for comparison between Lixisenatide vs Insulin glulisine TID in HbA1c and body weight. If both comparisons were met, then both would be declared significant. Otherwise, if only one was met, then the one met should be tested at α=0.0125 (1-sided); Test type: Non-Inferiority or Equivalence — Pre-specified non-inferiority margin of 0.4%; ANCOVA; LS Mean Difference = 0.21, 95% CI 2-sided [0.095 to 0.328], Standard Error of Mean 0.059 — Lixisenatide vs Insulin Glulisine TID

2. Primary Outcome: Change in Body Weight From Baseline to Week 26
Description: Primary outcome was the comparison between Lixisenatide versus Insulin Glulisine TID.
  Change in body weight was calculated by subtracting baseline value from Week 26 value. Missing data was imputed using LOCF. On-treatment period for this efficacy variable was defined as the time from the first dose of study drug up to 3 days after the last dose of study drug.
Time Frame: Baseline, Week 26
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline body weight assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 295 | 295 | 295
kg | -0.63 (0.276) | 1.03 (0.276) | 1.37 (0.271)
Statistical Analysis 1: Comparison: Lixisenatide vs Insulin Glulisine TID; Analysis was performed using ANCOVA model as described above. Hochberg procedure was used to control type 1 error at α = 0.025 (1-sided) for comparison between lixisenatide vs insulin glulisine TID in HbA1c and body weight. If both comparisons were met, then both would be declared significant. Otherwise, if only one was met, then the one met should be tested at α=0.0125 (1-sided); Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; The superiority was assessed by comparing the P-value at significance level = 0.025 or 0.0125; LS Mean Difference = -1.99, 95% CI 2-sided [-2.593 to -1.396], Standard Error of Mean 0.305 — Lixisenatide vs Insulin Glulisine TID

3. Secondary Outcome: Percentage of Participants With HbA1c Level <7% and ≤6.5% at Week 26
Description: The on-treatment period for this efficacy variable was defined as the time from the first dose of study drug up to 14 days after the last dose of study drug. Missing data was imputed using LOCF.
Time Frame: Week 26
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline HbA1c assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 292 | 292 | 295
percentage of participants
  HbA1c ≤6.5% | 20.5 | 17.8 | 30.8
  HbA1c <7.0% | 42.1 | 38.4 | 49.2

4. Secondary Outcome: Percentage of Participants With no Weight Gain at Week 26
Description: The on-treatment period for this efficacy variable was the time from the first dose of study drug up to 3 days after the last dose of study drug.
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 295 | 295 | 295
percentage of participants | 64.7 | 36.6 | 30.5

5. Secondary Outcome: Change in Average 7-point SMPG Profiles From Baseline to Week 26
Description: Participants recorded a 7-point plasma glucose profile measured before and 2 hours after each meal and at bedtime three times in a week before baseline, before visit Week 12 and before visit week 26 and the average value across the profiles performed in the week a visit for the 7-time points was calculated. Change in average 7-point SMPG was calculated by subtracting baseline value from Week 26 value. Missing data was imputed using LOCF. The on-treatment period for this efficacy variable was defined as the time from the first dose of study drug up to the day of last dose of study drug.
Time Frame: Baseline, Week 26
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline 7-point SMPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 270 | 268 | 278
mmol/L | -0.784 (0.1141) | -0.782 (0.1133) | -1.053 (0.1105)

6. Secondary Outcome: Change in FPG From Baseline to Week 26
Description: Change in FPG was calculated by subtracting baseline value from Week 26 value. Missing data was imputed using LOCF. The on-treatment period for this efficacy variable was the time from the first dose of study drug up to 1 day after the last dose of study drug.
Time Frame: Baseline, Week 26
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline FPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 295 | 295 | 294
mmol/L | -0.23 (0.143) | -0.21 (0.142) | -0.06 (0.14)

7. Secondary Outcome: Change in PPG From Baseline to Week 26 (in Participants Who Had an Injection of Investigational Medicinal Product [IMP] Before Breakfast)
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Change in PPG was calculated by subtracting baseline value from Week 26 value. Missing data was imputed using LOCF. The on-treatment period for this efficacy variable was the time from the first dose of study drug up to the day of last dose of study drug.
Time Frame: Baseline, Week 26
Population: mITT population. Here, number of participants analyzed = participants with IMP injection before breakfast and baseline and at least one post-baseline 2-hour PPG assessment during on-treatment period.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 69 | 55 | 68
mmol/L | -3.93 (4.29) | -1.62 (4.01) | -1.87 (3.18)

8. Secondary Outcome: Change in Glucose Excursions From Baseline to Week 26 (in Participants Who Had an Injection of IMP Before Breakfast)
Description: Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the standardized meal test, before study drug administration. Change in glucose excursions was calculated by subtracting baseline value from Week 26 value. Missing data was imputed using LOCF. The on-treatment period for this efficacy variable was the time from the first dose of study drug up to the day of last dose of study drug.
Time Frame: Baseline, Week 26
Population: mITT population. Here, number of participants analyzed = participants with IMP injection before breakfast and baseline and at least one post-baseline glucose excursion assessment during on-treatment period.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 64 | 53 | 66
mmol/L | -3.42 (4.13) | -1.59 (3.42) | -1.56 (2.52)

9. Secondary Outcome: Change in Insulin Glargine Dose From Baseline to Week 26
Description: Change in Insulin glargine dose was calculated by subtracting the baseline value from Week 26 value. Missing data was imputed using LOCF. The on-treatment period for this efficacy variable was the time from the first dose of study drug up to the day of last dose of study drug.
Time Frame: Baseline, Week 26
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline insulin glargine dose assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: U
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 292 | 294 | 294
U | 0.7 (1.002) | -0.06 (0.999) | -3.13 (0.982)

10. Secondary Outcome: Insulin Glulisine Dose at Week 26
Description: The on-treatment period for this efficacy variable was the time from the first dose of study drug up to the day of last dose of study drug. Missing data was imputed using LOCF.
Time Frame: Week 26
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline insulin glulisine dose assessment during on-treatment period.
Measure: Mean (Standard Deviation); unit: U
Arm/Group | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 295 | 293
U | 9.97 (7.8) | 20.24 (13.04)

11. Secondary Outcome: Total Insulin Dose at Week 26
Description: The on-treatment period for this efficacy variable was the time from the first dose of study drug up to the day of last dose of study drug. Missing data was imputed using LOCF.
  The outcome is reporting results of total insulin (amounts of Insulin Glargine plus Insulin Glulisine ) only for the arms in which Insulin Glulisine was administered and is not applicable for the lixisenatide arm in which only Insulin Glargine is administered. Change in dose of the insulin used by patients in the Lixisenatide arm (i.e. Insulin Glargine) is reported in the secondary Outcome Measure 9.
Time Frame: Week 26
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline total insulin dose assessment during on-treatment period.
Measure: Mean (Standard Deviation); unit: U
Arm/Group | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 295 | 294
U | 73.61 (39.13) | 81.05 (33.55)

12. Secondary Outcome: Percentage of Participants With Documented Symptomatic and Severe Symptomatic Hypoglycemia
Description: Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <60 mg/dL (3.3 mmol/L). Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the participant required the assistance of another person and was associated with either a plasma glucose level below 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose administration (maximum of 185 days)
Population: All randomized participants who were exposed to at least one dose of study drug, regardless of the amount of treatment administered.
  The 4 participants in the TID group who received Insulin Glulisine QD were analyzed according to the QD dose.The 1 participant in the QD group who received Insulin Glulisine TID was analyzed according to the TID dose
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 298 | 301 | 294
percentage of participants
  Documented symptomatic hypoglycemia | 31.5 | 37.5 | 44.6
  Severe symptomatic hypoglycemia | 0 | 0.7 | 0

13. Secondary Outcome: Percentage of Participants Who Reached the Target of HbA1c <7% at Week 26 and Did Not Experienced Documented (Plasma Glucose <60 mg/dL) Symptomatic Hypoglycemia During 26 Week Treatment Period
Description: The on-treatment period for HbA1c assessment was defined as the time from the first dose of study drug up to 14 days after the last dose of study drug. The on-treatment period for symptomatic hypoglycemia assessment was defined as the time from the first dose of study drug up to 1 day after the last dose of study drug.
Time Frame: Week 26
Population: mITT population. Participants without any post-baseline on-treatment value for HbA1c were counted as non-responders if they experienced at least one symptomatic hypoglycemia. Otherwise, they were counted as missing.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 296 | 293 | 295
percentage of participants | 29.4 | 24.2 | 26.1

14. Secondary Outcome: Percentage of Participants Who Reached the Target of HbA1c <7% and Had no Weight Gain at Week 26
Description: The on-treatment period for HbA1c assessment was defined as the time from the first dose of study drug up to 14 days after the last dose of study drug. The on-treatment period for body weight assessment was defined as the time from the first dose of study drug up to 3 days after the last dose of study drug.
Time Frame: Week 26
Population: mITT population. Participants without post-baseline on-treatment values (for HbA1c and body weight) that were no more than 30 days apart were counted as non-responders if at least one of the components (HbA1c and/or body weight) was available and showed non-response. Otherwise, they were counted as missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 295 | 293 | 295
percentage of participants | 31.2 | 16.7 | 17.6

15. Secondary Outcome: Percentage of Participants Who Reached the Target of HbA1c <7%, Had no Weight Gain at Week 26, and Did Not Experience Documented (Plasma Glucose <60 mg/dL) Symptomatic Hypoglycemia During 26-Week Treatment Period
Description: The on-treatment period for HbA1c assessment was defined as the time from the first dose of study drug up to 14 days after the last dose of study drug. The on-treatment period for body weight assessment was defined as the time from the first dose of study drug up to 3 days after the last dose of study drug. The on-treatment period for symptomatic hypoglycemia assessment was defined as the time from the first dose of study drug up to 1 day after the last dose of study drug. Participants without post-baseline on-treatment values (HbA1c and body weight) that were no more than 30 days apart were counted as non-responders if at least one of the components (HbA1c and/or body weight) was available and showed non-response, or if they experienced at least one documented symptomatic hypoglycemia during the on-treatment period. Otherwise, they were counted as missing data.
Time Frame: Week 26
Population: mITT population.Participants without post-baseline on-treatment values(HbA1c;body weight),no more than 30 days apart counted as non-responders if at least one of components(HbA1c;body weight) was available,showed non-response or experienced at least one symptomatic hypoglycemia during on-treatment period.Otherwise,they were counted as missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Number analyzed (Participants) | 297 | 294 | 295
percentage of participants | 22.2 | 9.2 | 10.8

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Day 185) regardless of seriousness or relationship to IMP.
Description: Reported AEs are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from the first dose of study drug up to 3 days after the last dose of study drug). Analysis was done on safety population.
  4 participants randomized to TID group, but received insulin glulisine QD were analyzed according to the QD dose. 1 participant randomized to QD group, but received insulin glulisine TID was analyzed according to the TID dose.
Groups:
- Lixisenatide: Lixisenatide 10 mcg QD SC for 2 weeks, then at a maintenance dose of 20 mcg QD up to Week 26 on top of insulin glargine with or without metformin (Median exposure of 182 days).
- Insulin Glulisine QD: Insulin glulisine QD SC up to Week 26 on top of Insulin glargine with or without metformin (Median exposure of 182 days).
- Insulin Glulisine TID: Insulin glulisine TID SC up to Week 26 on top of Insulin glargine with or without metformin (Median exposure of 182 days).
Arm/Group | Lixisenatide | Insulin Glulisine QD | Insulin Glulisine TID
Serious Adverse Events (participants affected / at risk) | 11/298 | 11/301 | 14/294
Other Adverse Events (participants affected / at risk) | 183/298 | 186/301 | 195/294
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide (N=298) | Insulin Glulisine QD (N=301) | Insulin Glulisine TID (N=294)
Erysipelas (Infections and infestations) | 1 | 0 | 0
Penile infection (Infections and infestations) | 1 | 0 | 0
Septic arthritis staphylococcal (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 2
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 | 2 | 0
Neuritis cranial (Nervous system disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hepatic mass (Hepatobiliary disorders) | 1 | 0 | 0
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 2 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide (N=298) | Insulin Glulisine QD (N=301) | Insulin Glulisine TID (N=294)
Nasopharyngitis (Infections and infestations) | 14 | 21 | 18
Hypoglycaemia (Metabolism and nutrition disorders) | 107 | 140 | 154
Headache (Nervous system disorders) | 20 | 8 | 12
Nausea (Gastrointestinal disorders) | 75 | 5 | 3
Vomiting (Gastrointestinal disorders) | 26 | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 20 | 10 | 4
Blood glucose decreased (Investigations) | 60 | 67 | 82
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 12 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.